CLINICAL TRIAL: NCT03793270
Title: Characterization of the Phenotypic Markers of B Cell Lymphocytes in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Rayan Mohammed, Principle investigator, Assiut University
Other Study IDs: 17200278
Record Dates: First submitted 2019-01-01; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Autoimmune Diseases
Keywords: Rheumatoid arthritis RA - B cells (B Lymphocyte).
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients: 1. Group 1: 30 diseased with Early Rheumatoid Arthritis from 6months to 1 year).
  drugs described in the clinic.
  Interventions: Diagnostic Test: for patients and healthy donors
- patients 2: 2. Group 2: 30 diseased with late/chronic Rheumatoid Arthritis. drugs described in the clinic.
  Interventions: Diagnostic Test: for patients and healthy donors
- healthy donors: 3. Group 3: 30 healthy controls. No drugs.
  Interventions: Diagnostic Test: for patients and healthy donors

INTERVENTIONS:
Diagnostic Test: for patients and healthy donors — 1. Detection of (CD19, CD24, CD38 & CD27) markers in peripheral blood samples by Flow Cytometry
  2. Determine the serum level of IL 10 using ELISA plate

SUMMARY:
Rheumatoid Arthritis (RA):

RA is a chronic inflammatory autoimmune disease that primarily affects the small joints, eventually leading to bone erosion and an inability to move (1). Several immune cells participate in the pathogenesis of RA. One of those cells is B cell.

DETAILED DESCRIPTION:
B cell population:

B lymphocytes play several critical roles in the pathogenesis of rheumatoid arthritis. They are the source of the rheumatoid factors (RF) and anti-cyclic-citrullinated peptide (anti-CCP), which contribute to immune complex formation and complement activation in the joints (2).

There is different B cell subpopulation according to the stage of maturation and activity. Distinction of this subpopulation can be done by detection of different CD molecules expressed on cell surface (3). From all sub-population this research will focus on these immunophenotypes; immature, mature, memory and B-reg cells by using CD 19, CD24, CD38 & CD27 respectively.

Joa˜ o E. Fonseca and his team found the reduction in B cell subpopulation especially (Pre- switched memory B cells) both in RA and Arthritis in the early stage. This observation not related to using methotrexate or corticosteroid in the treatment. They used the classification of B cells with CD 19 mainly and then IgD and CD27 to identify B cells (4).

Gabriella Sármay team found that the number of B-reg CD19+ CD27+ IL-10+ cells in peripheral blood is fewer in RA patients compared with healthy controls (5).

Interleukin 10:

Interleukin (IL)-10 functions as an anti-inflammatory cytokine in rheumatoid arthritis. IL-10 mRNA levels were significantly elevated in synovial fluid mononuclear cells (SFMCs) from patients with RA compared with PBMCs peripheral blood mononuclear cells (PBMCs) from RA patients or healthy volunteers according to Isomäki P (6).

IL 10 is primarily produced by monocytes mainly and, then by lymphocytes; type 2 T helper cells (TH2), mast cells, CD4+CD25+Foxp3+ regulatory T cells, and in a certain subset of activated T cells and B cells (7).

ELIGIBILITY:
Inclusion criteria:

* Patient diagnosed as Rheumatoid arthritis that fulfilled ACR/EULAR Criteria (American College of Rheumatology/European League Against Rheumatism).
* (8) Age >18 Years.

  b. Exclusion criteria:
* Diagnosed patients with other autoimmune disease or other infections.
* Pregnant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total sample size will be 90 samples will be divided into groups:
  1. Group 1: 30 diseased with Early Rheumatoid Arthritis from 6months to 1 year).
  2. Group 2: 30 diseased with late/chronic Rheumatoid Arthritis.
  3. Group 3: 30 healthy controls.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-03 (Estimated); Primary Completion 2019-08-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Detection of the percentage (%) B cell subpopulation in early-detected Rheumatic arthritis before taking long course medication and in late Rheumatic arthritis. Detection of the level of IL 10 in the serum for all patients. | after 6 monthes
  WBCs will be isolated from whole blood sample, then different monoclonal antibodies labeled with different markers will mixed with sample to be used for measuring the percent of each in the B cell population. Serum Samples will be collected and preserved in -80 degree then all samples will be measured with Elisa according to the manufacture procedures.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverman GJ, Carson DA. Roles of B cells in rheumatoid arthritis. Arthritis Res Ther. 2003;5 Suppl 4(Suppl 4):S1-6. doi: 10.1186/ar1010. Epub 2003 Dec 2. PMID 15180890